CLINICAL TRIAL: NCT04946344
Title: Cherokee Health for Elderly Residents With Osteoarthritis of the Knee in the Eastern Band
Brief Title: The Cherokee Study: Cherokee Health for Elderly Residents With Osteoarthritis of the Knee
Acronym: Cherokee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00033618 - Cherokee; U01AR068658 (NIH)
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis
Keywords: Knee Pain; Exercise; Diet; Weight Loss
MeSH Terms: conditions — Osteoarthritis; Motor Activity; Weight Loss | interventions — Diet; Exercise

STUDY DESIGN:
Intervention Model Description: 30 ambulatory, community-dwelling persons that meet the ACR clinical criteria for knee osteoarthritis
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet & Exercise (Experimental): Participants will attend an exercise class 3 days/week for 3 months. The exercise program will consist of a 15-minute aerobic phase, a 20-minute strength training phase, a second 15-minute aerobic phase, and a 10 minute cool down phase. Participant's will also attend individual and group diet sessions. Each participant will be prescribed an individual walking prescription by the exercise leader, which will be adjusted accordingly, as each participant progresses throughout the 3 months. The exercise will be of moderate intensity. Alternate forms of aerobic exercise, such as but not limited to stationary bike, elliptical trainer, or treadmill walking, can be used in place of over-ground walking. This choice could be based on participant preference, the limitations of the exercise facility, or the participant's pain level.
  Interventions: Behavioral: Diet & Exercise
- Attention Control (Active Comparator): The attention control intervention will cover an 3 month period. There will be two face to face group meetings over the 3 months, with one meeting each at months 1 and 3; and during the other months (month 2) participants will receive a combination of text messages, emails, and phone calls based on continued monitoring of participant needs and delivered via their preferred mode of contact.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Diet & Exercise — Participants will attend exercise and diet classes.
  Arms: Diet & Exercise
Behavioral: Attention Control — Participants will attend healthy living classes and receive phone calls/emails/texts.
  Arms: Attention Control

SUMMARY:
This study aims to develop and demonstrate the effectiveness of a systematic, practical, cost-effective diet-induced weight loss and exercise intervention in Cherokee, North Caroling that will recruit American Indian participants; that can reduce pain and improve other clinical outcomes in knee OA patients. This pragmatic community-based trial will determine if the investigators previous findings translate to real-world settings and will address common concerns about barriers to effectiveness/ implementation.

DETAILED DESCRIPTION:
Obesity is a modifiable risk factor for knee osteoarthritis (OA), and weight loss is an effective non-pharmacologic treatment to reduce pain. Recently, the investigators determined that under ideal, highly controlled circumstances, a diet-induced weight loss of 10% combined with exercise was significantly better at reducing pain than either intervention alone. Compared to the investigators previous longterm weight loss and exercise trials of knee OA, the diet-induced weight loss and exercise group was twice as effective at relieving pain. Whether the investigators results can be generalized to less rigorously monitored patient cohorts is unknown. Thus the challenge the investigators now face is to provide the practical means to implement this proven treatment in the community setting. This study aims to develop and demonstrate the effectiveness of a systematic, practical, cost-effective diet-induced weight loss and exercise intervention in both urban and rural communities that can reduce pain and improve other clinical outcomes in knee OA patients.

Participants will be 30 ambulatory, community-dwelling, overweight and obese men and women who meet the American College of Rheumatology clinical criteria for knee OA. The primary aim is to determine whether a pragmatic, community-based 3-month diet-induced weight loss and exercise intervention implemented in Cherokee, North Carolina significantly decreases knee pain in overweight and obese adults with knee OA relative to an attention control group. Secondary aims will determine whether this intervention improves self-reported function, health-related quality of life, and mobility. The investigators will also establish the cost-effectiveness of this pragmatic, community-based, multimodal diet-induced weight-loss and exercise program by conducting cost-effectiveness and budgetary impact analyses using data from the current trial in a validated computer-simulated model of knee OA.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 50
* Knee Pain plus American College of Radiology (ACR) Criteria for Knee Osteoarthritis
* BMI = 25 ≥ kg/m2

Exclusion Criteria:

* Significant co-morbid disease that would threaten safety or impair ability to participate in interventions or testing (Blindness; Type 1 diabetes; Severe coronary artery disease)
* Not sufficiently overweight or obese, BMI < 27 kg/m2
* Not having knee pain
* Inability to finish 3-month study or unlikely to be compliant (Planning to leave area > 1 month during the next 3 months; Unwilling to change eating or physical activity habits; Unwilling to discontinue pain medication use for 3 days prior to testing visit)
* Living > 30 minutes from the intervention site
* Age, age < 50
* Other conditions that may prohibit the effective delivery of the intervention (Unable to provide own transportation to exercise center; Unable to read or write)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Messier, PhD, Principal Investigator — Wake Forest University
Locations (2):
- United States (2):
  - Ginger Welch Complex, Cherokee, North Carolina
  - Wake Forest University/Wake Forest University Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
All of the individual data that has been collected during the trial after it has been deidentified will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available 6 months after study analysis has been completed.
Access Criteria: Persons wishing to receive data must submit a formal request to the study team. Consultation with the leaders of tribe is required and approval must be given prior to data access.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diet & Exercise | Attention Control
Started | 8 | 8
Completed | 6 | 6
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diet & Exercise | Attention Control | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (8.7) | 66.5 (8.3) | 65.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 5 | 9
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34.7 (7.7) | 32.5 (6) | 33.6 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario McMasters Universities Osteoarthritis Index (WOMAC) - Knee Pain
Description: Western Ontario McMasters Universities Osteoarthritis Index (WOMAC) pain subscale in overweight and obese adults with knee OA compared to an attention-control group - The pain index assesses participants' pain on the same scale, ranging from 0 (none) to 4 (extreme). The pain subscale consists of 5 items. Normalized values are reported. To calculate, the mean score of the individual items of is divided by 4 (the highest possible score for a single answer option). The mean of the observed items is then multiplied by 100 and subtracted from 100. Total scores can range from 0-100, with larger scores indicating greater pain.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diet & Exercise | Attention Control
Number analyzed (Participants) | 6 | 6
score on a scale | 67.13 (19.86) | 62.04 (25.79)

2. Secondary Outcome: Western Ontario McMasters Universities Osteoarthritis Index (WOMAC) - Function
Description: Western Ontario McMasters Universities Osteoarthritis Index (WOMAC) function subscale in overweight and obese adults with knee OA compared to an attention-control group - participants indicate on a scale from 0 (none) to 4 (extreme) the degree of difficulty experienced in the last week due to knee OA. Scores range from 0 to 96 for the total WOMAC where 0 represents the best health status and 96 the worst possible status. The higher the score, the poorer the function.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diet & Exercise | Attention Control
Number analyzed (Participants) | 6 | 6
score on a scale | 74.10 (21.18) | 66.16 (14.43)

3. Secondary Outcome: Health Related Quality of Life (SF-36)
Description: The physical dimension of the SF-36 is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. A higher score represents a more favorable health state.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diet & Exercise | Attention Control
Number analyzed (Participants) | 6 | 6
score on a scale | 42.20 (31.11) | 31.32 (22.71)

4. Secondary Outcome: Distance Walked - Mobility (Six Minute Walk)
Description: To determine whether a pragmatic, community-based, 3-month, diet-induced weight-loss and exercise intervention improves 6-minute walk distance (an accepted measure of mobility) in overweight and obese adults with knee OA compared to an attention control group.
Time Frame: Month 3
Population: Number of participants is reduced as some subjects opted to not return for in person testing.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Diet & Exercise | Attention Control
Number analyzed (Participants) | 2 | 2
meters | 431.9 (87.5) | 296.9 (252.2)

5. Other Pre Specified Outcome: Physical Performance Battery (SPPB) - Balance
Description: A score lower than 10 indicates one or more mobility limitations. A score lower than 10 is predictive of all-cause mortality
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Physical Performance Battery (SPPB) - Walking Speed
Description: as for outcome 5
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Physical Performance Battery (SPPB) - Chair Rise
Description: as for outcome 5
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Physical Performance Battery (SPPB) - Stair Activity
Description: Ascending and descending stair activity measured by the time (in seconds) it takes to ascend and descend a flight of 8 steps with 20cm (8 inch) step height
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

9. Other Pre Specified Outcome: EuroQol Quality of Life
Description: Evaluates the generic quality of life developed in Europe and widely used. The EuroQol Quality (EQ)-five dimensions (5D) descriptive system is a preference-based Health-related quality of life (HRQL) measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

10. Other Pre Specified Outcome: The Walking Efficacy for Duration Scale
Description: Duration is a measure to determine participants' beliefs in their physical capability to successfully complete incremental 5-minute intervals (5 to 40 minutes) at a moderately fast pace For each item, participants indicate their confidence to execute the behavior on a 100-point percentage scale comprised of 10-point increments, ranging from 0% (not at all confident) to 100% (highly confident). Total strength for each measure of self-efficacy is then calculated by summing the confidence ratings and dividing by the total number of items in the scale, resulting in a maximum possible efficacy score of 100
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

11. Other Pre Specified Outcome: The Positive and Negative Affect (PANAS)
Description: Measures both positive and negative affect, leading to more insightful outlooks regarding participants' feeling states. This scale consists of 20 items that reflect the intensity of how the participant "feels" right now
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

12. Other Pre Specified Outcome: The Gait Efficacy/Environmental Efficacy Scale
Description: Will ask the participants' confidence in performing certain activities
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Satisfaction With Life Scale
Description: Focused to assess global life satisfaction - Participants indicate how much they agree or disagree with each of the 5 items using a 7-point scale that ranges from 7 strongly agree to 1 strongly disagree
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

14. Other Pre Specified Outcome: The Weight Efficacy Lifestyle Questionnaire (WEL)
Description: A 20-item measure employed to assess self-efficacy for weight management - 10-point Likert scale ranging from 0 (not confident) to 9 (very confident) to resist the desire to eat.
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

15. Other Pre Specified Outcome: The Perceived Stress Scale (PSS)
Description: Will measure the degree to which people perceive their lives as stressful - PSS-10 scores are obtained by reversing the scores on the four positive items: For example, 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4, 5, 7, and 8 are the positively stated items. Scores around 13 are considered average. Higher scores indicate higher stress.
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

16. Other Pre Specified Outcome: The Adherence Self-efficacy Questionnaire
Description: Assess beliefs in one's ability (confidence) to continue exercising at various intensities and frequencies - This 12-item scale assessed patient confidence to carry out important treatment-related behaviors related to adhering to treatment plans, including medication regimen adherence and following plans for nutrition, exercise, etc, in the face of barriers - Higher scores indicate a greater level of self-efficacy
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Pain Catastrophizing Scale (PCS)
Description: People are asked to indicate the degree to which they have the above thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale. A total score is yielded (ranging from 0-52), along with three subscale scores assessing rumination, magnification and helplessness
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The KOOS questionnaire will be used to assess the patient's opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury and also consequences of primary osteoarthritis (OA) - the mean score of the individual items of each subscale and divide by 4 (the highest possible score for a single answer option). Traditionally in orthopedics, 100 indicates no problems and 0 indicates extreme problems
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Intermittent and Constant Osteoarthritis Pain (ICOAP)
Description: The ICOAP assesses pain in individuals with knee osteoarthritis taking into account both constant and intermittent pain experiences - the 11 items are scored from 0-4 with 0 being no pain and 4 being extreme pain - maximum score = 100
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

20. Other Pre Specified Outcome: (DHQ) Dietary History Questionnaire
Description: The diet history method is a detailed retrospective dietary assessment which obtains details of individual foods, and comprehensive information about foods eaten less regularly
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Behavioral Risk Factor Surveillance System (BRFSS)
Description: The BRFSS is a cross-sectional telephone survey that measures health literacy - the nation's premier system of health-related telephone surveys that collect state data about U.S. residents regarding their health-related risk behaviors, chronic health conditions, and use of preventive services.
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

22. Other Pre Specified Outcome: The Physical Activity Scale for the Elderly (PASE)
Description: The PASE assesses the types of activities typically chosen by older adults (walking, recreational activities, exercise, housework, yard work, and caring for others. It uses frequency, duration, and intensity level of activity over the previous week to assign a score, ranging from 0 to 793, with higher scores indicating greater physical activity -Total PASE scores are computed by multiplying activity weights by activity frequencies
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

23. Other Pre Specified Outcome: The Montreal Cognitive Assessment (MOCA)
Description: During the MOCA, a health professional asks a patient a series of questions designed to test a range of everyday mental skills. The maximum MOCA score is 30 points. A score of 20 to 24 suggests mild dementia, 13 to 20 suggests moderate dementia, and less than 12 indicates severe dementia
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Center for Epidemiologic Studies Depression Scale
Description: The score is the sum of the 20 questions. Possible range is 0-60. If more than four questions are missing answers, do not score the Center for Epidemiologic Studies Depression (CES-D) questionnaire. A score of 16 points or more is considered depressed
Time Frame: Baseline and Month 3
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Cost-effectiveness
Description: Resource utilization will be collected by questionnaire, with domains including visits to clinicians (physicians, nurses, physical therapists, others), tests, medications, injections, surgery, alternative therapies. The Work Productivity and Activity Impairment index (WPAI) will be used to assess absenteeism and reduced productivity while at work
Time Frame: Month 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Diet & Exercise | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT04946344/Prot_001.pdf
  • Informed Consent Form (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT04946344/ICF_000.pdf